CLINICAL TRIAL: NCT03907293
Title: Effect of a Cardiac Rehabilitation (CR) Programme on Protein Molecules Associated With Arterial Function, and an Exploration of Reasons for Agreeing or Declining to Participate in a CR Programme
Brief Title: Effect of a Cardiac Rehabilitation (CR) Programme on Molecular Mechanisms
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other); South Eastern Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0056
Record Dates: First submitted 2019-03-19; First posted 2019-04-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis; Myocardial Infarction; Myocardial Ischemia
Keywords: Cardiac Rehabilitation; Exercise; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Myocardial Ischemia; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Whole blood Lymphocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase-III Cardiac Rehabilitation: Eight weeks of supervised exercise sessions (one session per week).
  Interventions: Behavioral: Exercise-based cardiac rehabilitation
- Phase-III and Phase IV Cardiac Rehabilitation: Twenty weeks of supervised exercise sessions (one session per week for first eight weeks [phase-III], session frequency determined by participant for remaining twelve weeks [phase-IV].
  Interventions: Behavioral: Exercise-based cardiac rehabilitation
- No Cardiac Rehabilitation: Participants who declined to take part in a cardiac rehabilitation programme.

INTERVENTIONS:
Behavioral: Exercise-based cardiac rehabilitation — Moderate intensity aerobic exercise, lifestyle advice, and psychological support.
  Groups: Phase-III Cardiac Rehabilitation; Phase-III and Phase IV Cardiac Rehabilitation

SUMMARY:
This study will evaluate the effect of a cardiac rehabilitation (CR) programme on blood protein molecules that may improve the function of arteries in coronary artery disease (CAD) patients who have suffered a heart attack. CAD patients who have either agreed or disagreed to take part in a CR programme will be recruited. This will allow a comparison of the study measurements between a group of patients who complete a CR programme and a group of patients who do not.

The other objective of this study is to perform interviews with the study participants and their significant others (i.e. spouse, family member, or a close friend) to listen to the reasons why patients agreed or disagreed to take part in a CR programme.

DETAILED DESCRIPTION:
An exercise-based cardiac rehabilitation (CR) programme is an established method of secondary prevention of coronary artery disease (CAD). Moreover, there is a body of evidence that supports the ability of this intervention to reduce hospital readmissions and cardiovascular mortality. However, despite the proven benefit, CR programmes are underutilised worldwide. Moreover, the molecular mechanisms responsible for orchestrating the beneficial physiological adaptations induced by a CR programme are poorly understood.

Therefore, this study will evaluate the effect of a CR programme on novel molecular mechanisms and endothelial function in post-myocardial infarction CAD patients. Additionally, semi-structured interviews will be conducted with study participants and their significant others (i.e. spouse, family member, or a close friend) to explore the reasons why patients may agree or disagree to take part in a CR programme. Altogether, this study will provide physiological and detailed qualitative information that may help to provoke an increased participation in CR programmes.

ELIGIBILITY:
Inclusion Criteria:

* Formally diagnosed coronary artery disease with evidence of ST- elevated or non-ST elevated myocardial infarction, as determined by evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia, and the detection of a rise and / or fall in cardiac biomarker values (preferably cardiac troponin), with at least one value above the 99th percentile upper reference limit, along with at least one of the following:

Symptoms of ischaemia, such as: extreme fatigue, breathlessness, chest pain, and heart palpitations.

New or presumed new significant ST-segment-T wave changes or new left bundle branch block.

Development of pathological Q waves on the electrocardiogram.

Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Identification of an intracoronary thrombus by angiography

* Over 18 years of age.
* Male or Female.
* Provision of informed consent.
* Ability to speak and write in English.
* Patients who have agreed to participate in a phase-III cardiac rehabilitation programme must be willing to attend the supervised group exercise sessions.
* No hospital readmissions with unstable symptoms (e.g. chest pain, shortness of breath, discomfort, or nausea) during the previous 4-weeks.
* Willing to comply with trial requirements.

Exclusion Criteria:

* Unstable angina pectoris (angina at rest or persistent angina regardless of pharmacological treatment e.g. glyceryl trinitrate).
* Uncontrolled cardiac arrhythmia.
* Survivor of cardiac arrest or cardiogenic shock.
* Any form of anaemia (haemoglobin < 90 grams / litre).
* Hepatic failure.
* Uncontrolled hypertension (resting systolic measurement > 180 mm Hg and / or diastolic measurement > 100 mm Hg).
* History of Raynaud's phenomenon.
* Congenital or acquired physical abnormalities of both arms.
* Consumption of vitamins, herbal, testosterone, estrogen/ progesterone, or antioxidant supplementation.
* Pregnant.
* History of or diagnosed with any form of cancer.
* Current participation in a different research study.

Patient Inclusion Criteria for Interview Component of Study:

* Patient has either declined or agreed to participate in a phase-III or phase-IV cardiac rehabilitation programme.
* Sufficient English language skills to understand and participate in an interview discussion.
* Over 18 years of age.
* Identified significant other provides informed consent to participate in the study.

Patient Exclusion Criteria for Interview Component of Study:

- Identified significant other refuses to participate or provide informed consent.

Significant Other Inclusion Criteria for Interview Component of Study:

* Nominated by the patient and willing to participate.
* Impacted or involved throughout the period of the patient's cardiovascular complication and recovery (e.g. familial relation, co-habitant, or close-relationship).
* Sufficient English language skills to understand and participate in an interview discussion.
* Over 18 years of age.
* Patient provides informed consent to participate in the study.

Significant Other Exclusion Criteria for Interview Component of Study:

- Patient refuses to participate or provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post-myocardial infarction coronary artery disease patients who have been invited to participate in a phase-III cardiac rehabilitation programme with the Belfast Health and Social Care Trust or South Eastern Health and Social Care Trust.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Sirtuin 1 serum protein concentration | At baseline and after 22-weeks
  Measured in ng/mL

SECONDARY OUTCOMES:
Interleukin-6 serum protein concentration | Baseline, week-8, and week-22
  Measured in pg/mL
Interleukin-10 serum protein concentration | Baseline, week-8, and week-22
  Measured in pg/mL
Sirtuin 1 messenger ribonucleic acid gene expression | Baseline, week-8, and week-22
Interleukin-6 messenger ribonucleic acid gene expression | Baseline, week-8, and week-22
Interleukin-10 messenger ribonucleic acid gene expression | Baseline, week-8, and week-22
Erythrocyte sedimentation rate | Baseline, week-8, and week-22
  Millimetres per hour
Serum low-density lipoprotein value | Baseline, week-8, and week-22
Serum total cholesterol value | Baseline, week-8, and week-22
Serum triglyceride value | Baseline, week-8, and week-22
Serum high-density lipoprotein value | Baseline, week-8, and week-22
Lipid soluble antioxidants concentrations | Baseline, week-8, and week-22
Lipid hydroperoxide concentration | Baseline, week-8, and week-22
Ascorbyl free radicle concentration | Baseline, week-8, and week-22
Brachial flow-mediated dilatation | Baseline, week-8, and week-22
  Percentage increase in arterial diameter
Arterial stiffness (finger photo-plethysmography technique) | Baseline, week-8, and week-22
  Stiffness index
Incremental Shuttle Walk Test | Baseline, week-8, and week-22
  Distance walked (metres)
Systolic and diastolic blood pressure | Baseline, week-8, and week-22
  Millimetre of mercury
Resting heart rate | Baseline, week-8, and week-22
  Beats per minute
Body mass index | Baseline, week-8, and week-22
  Kilograms per metre squared
Waist circumference | Baseline, week-8, and week-22
  Centimetres

OTHER OUTCOMES:
Qualitative perspectives from study participants and their significant others regarding reasons for agreeing or declining to participate in a phase-III or phase-IV cardiac rehabilitation programme | Week-8 or week-22
  Generated by semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Hughes, PhD, Study Director — Ulster University; Gareth Thompson, PhD student, Study Chair — Ulster University; Gareth Davison, PhD, Study Chair — Ulster University; Jacqui Crawford, BSc, MSc, Study Chair — Ulster University; Lisa Spratt, Principal Investigator — Belfast Health and Social Care Trust; Maureen Morrison, Principal Investigator — South Eastern Health and Social Care Trust
Locations (2):
- United Kingdom (2):
  - Belfast Health and Social Care Trust (Belfast City Hospital, Mater Hospital, and Royal Victoria Hospital), Belfast, Co. Antrim
  - South Eastern Health and Social Care Trust (Ulster Hospital), Dundonald, Co. Down

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thompson G, Wilson IM, Davison GW, Crawford J, Hughes CM. "Why would you not listen? It is like being given the winning lottery numbers and deciding not to take them": semi-structured interviews with post-acute myocardial infarction patients and their significant others exploring factors that influence participation in cardiac rehabilitation and long-term exercise training. Disabil Rehabil. 2022 Aug;44(17):4750-4760. doi: 10.1080/09638288.2021.1919213. Epub 2021 May 7. PMID 33961501